CLINICAL TRIAL: NCT05189808
Title: Radiofrequency Ablation for Indeterminate Bethesda III Thyroid Nodules
Brief Title: Radiofrequency Ablation for BIII Thyroid Nodules
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jennifer Kuo, Associate Professor, Columbia University
Other Study IDs: AAAT1979
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Indeterminate Bethesda III Thyroid Nodules
Keywords: Radiofrequency Ablation
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Ultrasound guided radiofrequency ablation (non-experimental)

SUMMARY:
The purpose of this observational chart review study is to evaluate the efficacy and safety of Radiofrequency Ablation (RFA) for treatment of indeterminate thyroid nodules before and after RFA procedure. This is a data collection study in which the investigators ask patients to give access to information generated before and after RFA treatment of their condition. The RFA procedure uses image guidance to place an electrode through the skin into the target area. In RFA, high-frequency electrical currents are passed through an electrode, creating a small region of heat to treat the lesion.

DETAILED DESCRIPTION:
In the United States, there is an estimated 10% lifetime probability for developing a thyroid nodule.

Up to 15% of these nodules will prove to be malignant. The incidence of thyroid cancer is increasing and is the third leading cause of cancer in women; accordingly, identification of a nodule

1 cm or larger in diameter often prompts a sophisticated diagnostic evaluation comprised of sonographic pattern risk assessment combined with fine needle aspiration biopsy (FNAB), which enables the assessment of cellular morphologic features that could not be identified by means of clinical assessment or imaging. Ultrasound-guided FNAB has been shown to accurately classify 62-85% of thyroid nodules as benign, thereby avoiding diagnostic surgery. Yet, 20-30% of aspirations still yield indeterminate cytologic findings: "atypia (or follicular lesion) of undetermined significance," "follicular neoplasm or suspicious for follicular neoplasm," and "suspicious for malignancy with a risk of malignancy ranging from 6-75%." Most patients with cytologically indeterminate nodules are referred for diagnostic thyroid surgery, but the majority prove to have benign disease. For these patients, thyroid surgery is unnecessary, yet it exposes them to 2-10% risk of serious surgical complications, and most would require thyroid hormone replacement therapy for life. Research in recent years has focused on the potential of molecular diagnostic approaches that could capitalize on increasing knowledge of the molecular etiology of thyroid nodules and the transcriptional and mutation landscape of thyroid cancers to augment diagnostic accuracy of FNABs. Most molecular profiling tests demonstrate a high sensitivity and negative predictive value that helps to decrease the number of benign nodules undergoing unnecessary diagnostic surgery. However, these classified benign nodules may continue to grow and ultimately may need to undergo surgery due to compressive symptoms. Although thyroid surgery has always been the mainstay of treatment for symptomatic nodular goiters, and is associated with excellent outcomes in experienced hands, thyroid surgery carries a low risk of complications that include recurrent or superior laryngeal nerve injury leading to voice changes, hypoparathyroidism, hypothyroidism with need for thyroid hormone supplementation, and unsightly scarring. Although many patients with thyroid cancers find these risks acceptable, these risks are sometimes less acceptable to patients with benign disease. In an era when the medical field is treating thyroid diseases less aggressively, there is a pressing need to identify approaches to treat indolent malignant disease less invasively.

Introduced in the early 2000s, ultrasound-guided percutaneous ablation of thyroid lesions has emerged as a potential alternative to surgery in patients with benign thyroid nodules. Of the myriad ablation methods, the most commonly used technique is radiofrequency ablation (RFA). An expanding body of evidence shows that radiofrequency ablation and other percutaneous interventions are effective treatments for benign solid thyroid nodules, toxic adenomas, and thyroid cysts resulting in overall volume reduction ranges of 40-70% with durable resolution of compressive and hyperthyroid symptoms. In addition, RFA has been used as an effective alternative treatment in the management of locally recurrent thyroid cancers in patients who are not good surgical candidates. Although these percutaneous techniques have been steadily.

gaining acceptance in Europe and Asia over the past 20 years, they have been slow to be adopted in the US. There remains a dearth of data regarding clinical experience in the United States and no randomized clinical trials have been performed evaluating RFA vs active surveillance for micropapillary carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Indeterminate Bethesda III nodules that have been molecularly profiled benign with either Afirma Genomic Sequencing Classifier (GSC) or ThyroSeq v3 tests

Exclusion Criteria:

* cardiac arrthymias
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (>/= 18 years) who have biopsy proven indeterminate thyroid nodules (Bethesda III only) that have been molecular profiled benign, who refuse to undergo or are not good candidates for surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Nodule Volume | 12 months
  ((Volume (baseline) - Volume (12m))/Volume(baseline))*100

SECONDARY OUTCOMES:
Complications | 12 months
  Incidence of procedural complications including but not limited to infection, bleeding, voice change, nerve damage

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Kuo, MD MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durante C, Costante G, Lucisano G, Bruno R, Meringolo D, Paciaroni A, Puxeddu E, Torlontano M, Tumino S, Attard M, Lamartina L, Nicolucci A, Filetti S. The natural history of benign thyroid nodules. JAMA. 2015 Mar 3;313(9):926-35. doi: 10.1001/jama.2015.0956. PMID 25734734
- [Background] de Rienzo-Madero B, Sabra JP, Gand E, Donatini G, Kraimps JL. Unilateral benign multinodular versus solitary goiter: Long-term contralateral reoperation rates after lobectomy. Surgery. 2019 Jan;165(1):75-79. doi: 10.1016/j.surg.2018.04.074. Epub 2018 Nov 8. PMID 30415868
- [Background] Kim YS, Rhim H, Tae K, Park DW, Kim ST. Radiofrequency ablation of benign cold thyroid nodules: initial clinical experience. Thyroid. 2006 Apr;16(4):361-7. doi: 10.1089/thy.2006.16.361. PMID 16646682
- [Background] Na DG, Lee JH, Jung SL, Kim JH, Sung JY, Shin JH, Kim EK, Lee JH, Kim DW, Park JS, Kim KS, Baek SM, Lee Y, Chong S, Sim JS, Huh JY, Bae JI, Kim KT, Han SY, Bae MY, Kim YS, Baek JH; Korean Society of Thyroid Radiology (KSThR); Korean Society of Radiology. Radiofrequency ablation of benign thyroid nodules and recurrent thyroid cancers: consensus statement and recommendations. Korean J Radiol. 2012 Mar-Apr;13(2):117-25. doi: 10.3348/kjr.2012.13.2.117. Epub 2012 Mar 7. PMID 22438678
- [Background] Kim JH, Baek JH, Lim HK, Ahn HS, Baek SM, Choi YJ, Choi YJ, Chung SR, Ha EJ, Hahn SY, Jung SL, Kim DS, Kim SJ, Kim YK, Lee CY, Lee JH, Lee KH, Lee YH, Park JS, Park H, Shin JH, Suh CH, Sung JY, Sim JS, Youn I, Choi M, Na DG; Guideline Committee for the Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. 2017 Thyroid Radiofrequency Ablation Guideline: Korean Society of Thyroid Radiology. Korean J Radiol. 2018 Jul-Aug;19(4):632-655. doi: 10.3348/kjr.2018.19.4.632. Epub 2018 Jun 14. PMID 29962870
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Jeong WK, Baek JH, Rhim H, Kim YS, Kwak MS, Jeong HJ, Lee D. Radiofrequency ablation of benign thyroid nodules: safety and imaging follow-up in 236 patients. Eur Radiol. 2008 Jun;18(6):1244-50. doi: 10.1007/s00330-008-0880-6. Epub 2008 Feb 20. PMID 18286289
- [Background] Baek JH, Kim YS, Lee D, Huh JY, Lee JH. Benign predominantly solid thyroid nodules: prospective study of efficacy of sonographically guided radiofrequency ablation versus control condition. AJR Am J Roentgenol. 2010 Apr;194(4):1137-42. doi: 10.2214/AJR.09.3372. PMID 20308523
- [Background] Watt T, Barbesino G, Bjorner JB, Bonnema SJ, Bukvic B, Drummond R, Groenvold M, Hegedus L, Kantzer V, Lasch KE, Marcocci C, Mishra A, Netea-Maier R, Ekker M, Paunovic I, Quinn TJ, Rasmussen AK, Russell A, Sabaretnam M, Smit J, Torring O, Zivaljevic V, Feldt-Rasmussen U. Cross-cultural validity of the thyroid-specific quality-of-life patient-reported outcome measure, ThyPRO. Qual Life Res. 2015 Mar;24(3):769-80. doi: 10.1007/s11136-014-0798-1. Epub 2014 Sep 7. PMID 25194574
- [Background] Dobnig H, Amrein K. Monopolar Radiofrequency Ablation of Thyroid Nodules: A Prospective Austrian Single-Center Study. Thyroid. 2018 Apr;28(4):472-480. doi: 10.1089/thy.2017.0547. Epub 2018 Mar 20. PMID 29490593